CLINICAL TRIAL: NCT04080258
Title: Effectiveness of Osteopathic Manipulative Therapy in Paediatric Patients, With High Frequency Headache.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Antonio Francesco Urbino (Other)
Collaborators: Scuola Superiore di Osteopatia Italiana (Other)
Responsible Party: Sponsor-Investigator, Antonio Francesco Urbino, Director Pediatric Department, A.O.U. Città della Salute e della Scienza
Organization: A.O.U. Città della Salute e della Scienza (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0063257
Record Dates: First submitted 2019-09-04; First posted 2019-09-06 (Actual); Last update posted 2019-09-16 (Actual); Status verified 2019-09

CONDITIONS: Headache Disorders; Primary Headache Disorder
Keywords: Headache Disorders; Primary Headache
MeSH Terms: conditions — Headache Disorders; Headache Disorders, Primary | interventions — Manipulation, Osteopathic

STUDY DESIGN:
Intervention Model Description: A two arms randomized controlled trial. The experimental group will receive Osteopathic Manipulative Therapy and the Active Comparator will receive Light Touch Therapy.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The subjects will be randomly assigned to two groups, OMTh and LTT, and will be randomized from a computer-generated list prepared in advance by an external statistician. Allocation will be concealed with opaque sealed envelopes which will be opened after enrolment.
  The paediatrician in charge of the outcome assessor will be blinded to allocation concealment. The nurse staff, and the osteopath in charge of collecting the data will be blinded to group assignment.
  The two osteopaths in charge of Osteopathic Manipulative Therapy and Light Touch Therapy will be unblinded to group assignment.
  Data export will be performed by the external statistician. The blind-to-treatment allocation was tested using a post-treatment single question survey conducted by the pediatrician.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Osteopathic Manipulative Therapy (Experimental): Osteopathic Manipulative Therapy (OMTh). Patients in the OMTh group will receive 5 Osteopathic manipulative therapies: the first at baseline, the second after 1 week, the third after 3 weeks, and then 2 more treatments on a monthly basis. The protocol will last for three months.
  Interventions: Other: Osteopathic manipulative therapy (OMTh)
- Light Touch Therapy (Sham Comparator): Participants to the LTT group will receive the protocol at the same date of the OMTh group.
  Interventions: Other: Light Touch Therapy (LTT)

INTERVENTIONS:
Other: Osteopathic manipulative therapy (OMTh) — The Osteopathic Manipulative Therapy includes both evaluation and treatment. The evaluation is semi-structured, two osteopaths will assess the presence of somatic dysfunctions which have to include the hyoid-pharyngeal, laryngeal, temporo-mandibular and lingual areas.
  The therapy is based on the treatment of somatic dysfunctions with different approaches that include: the balanced ligamentous tension technique, the myofascial release, the visceral manipulation, and the balanced membranous tension technique. The OMTh lasts for 45 minutes of which 15 of evaluation and 30 of treatment.
  Arms: Osteopathic Manipulative Therapy
Other: Light Touch Therapy (LTT) — The Light Touch Therapy is a sham treatment consistent with the OMTh one during the phase of evaluation. The treatment retains the same areas used for osteopathic approach but avoids prolonged touch in any area of the body by moving the hands every few seconds and by flattening and softening the surface of the hands in order to minimize focal areas of force.
  Arms: Light Touch Therapy

SUMMARY:
The aim of this study is to evaluate the effectiveness of osteopathic manipulative therapy, in supporting prophylactic medications in paediatric patients, with high frequency headache.

DETAILED DESCRIPTION:
Headache is one of the most common medical complaints in childhood, with migraine and tension-type headaches (TTHs) being the most frequent diseases. The prevalence of tension-type headache (TTH) varies from 10% to 25% in school children and adolescents. Therefore a range varying from 0,1% to 5,9% of this population presents chronic tension-type headache, occuring at least 15 days on a monthly basis.

The tension-type headache is most likely multifactorial. In children, a connection seems possible between tension-type headache and psychosocial stress, psychiatric disorders, muscular stress, or oromandibular dysfunction.

The treatment of tension-type headache covers a systemic approach that includes both pharmacologic and nonpharmacologic therapies, such as biobehavioural management, and patient and family education regarding lifestyle modifications to develop and/or maintain healthy habits. Efficacy of these therapies is still unclear. Complementary therapies could be a good support to pharmacologic treatment. Osteopathic treatment results effective in some paediatric conditions, but in primary headache the possible efficacy is still unknown.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of primary high-frequency headache attacks.
* No reduction or inconsistent reduction of attacks after two months of prophylactic treatment.

Exclusion Criteria:

Secondary headache.

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 90 (Estimated)
Dates: Start 2018-06-18 (Actual); Primary Completion 2020-06-18 (Estimated); Study Completion 2020-12-18 (Estimated)

PRIMARY OUTCOMES:
Number of days with headache | At baseline (T0), after 1 month (T1), at 3 months from baseline (T2) and follow-up at 6 months from baseline.
  Difference in number of days per month with headache

SECONDARY OUTCOMES:
Reduction of analgesic use | At baseline (T0), after 1 month (T1), at 3 months form baseline (T2) and follow-up at 6 months from baseline
  Difference in reduction of analgesic use per month
Reduction of functional disability (school and leisure activity) | At baseline (T0), after 1 month (T1), at 3 months form baseline (T2) and follow-up at 6 months from baseline
  Days per month with functional disability.
Reduction of headache intensity | At baseline (T0), after 1 month (T1), at 3 months form baseline (T2) and follow-up at 6 months from baseline
  Difference in intensity of pain: mild, moderate and severe
Adverse event | From first treatment (1 week post-baseline) up to end of treatment course (3 months).
  Symptoms such as increased of pain that could occur after the Osteopathic Manipulative Therapy or Light Touch Therapy

CONTACTS AND LOCATIONS:
Overall Officials: Antonio F Urbino, Medical, Principal Investigator — A.O.U. Città della Salute e della Scienza
Locations (1):
- Centro Cefalee dell'età evolutiva - Ospedale Infantile Regina Margherita S.C. Pediatria d'Urgenza., Torino, Italy

REFERENCES:
- [Background] Huguet A, Tougas ME, Hayden J, McGrath PJ, Chambers CT, Stinson JN, Wozney L. Systematic Review of Childhood and Adolescent Risk and Prognostic Factors for Recurrent Headaches. J Pain. 2016 Aug;17(8):855-873.e8. doi: 10.1016/j.jpain.2016.03.010. Epub 2016 Apr 19. PMID 27102894
- [Background] Gofshteyn JS, Stephenson DJ. Diagnosis and Management of Childhood Headache. Curr Probl Pediatr Adolesc Health Care. 2016 Feb;46(2):36-51. doi: 10.1016/j.cppeds.2015.11.003. Epub 2015 Dec 29. PMID 26750538
- [Background] Kroon Van Diest AM, Powers SW. Cognitive Behavioral Therapy for Pediatric Headache and Migraine: Why to Prescribe and What New Research Is Critical for Advancing Integrated Biobehavioral Care. Headache. 2019 Feb;59(2):289-297. doi: 10.1111/head.13438. Epub 2018 Nov 16. PMID 30444269
- [Background] Posadzki P, Lee MS, Ernst E. Osteopathic manipulative treatment for pediatric conditions: a systematic review. Pediatrics. 2013 Jul;132(1):140-52. doi: 10.1542/peds.2012-3959. Epub 2013 Jun 17. PMID 23776117
- [Background] Cerritelli F, Ginevri L, Messi G, Caprari E, Di Vincenzo M, Renzetti C, Cozzolino V, Barlafante G, Foschi N, Provinciali L. Clinical effectiveness of osteopathic treatment in chronic migraine: 3-Armed randomized controlled trial. Complement Ther Med. 2015 Apr;23(2):149-56. doi: 10.1016/j.ctim.2015.01.011. Epub 2015 Jan 21. PMID 25847552